CLINICAL TRIAL: NCT05283109
Title: ETAPA I: Evaluation of Tumor Associated P30-Peptide Antigen I; A Pilot Trial of Peptide-based Tumor Associated Antigen Vaccines in Newly Diagnosed, Unmethylated, and Untreated Glioblastoma (GBM)
Brief Title: ETAPA I: Peptide-based Tumor Associated Antigen Vaccine in GBM
Acronym: ETAPA I
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mustafa Khasraw, MBChB, MD, FRCP, FRACP (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Mustafa Khasraw, MBChB, MD, FRCP, FRACP, Professor of Neurosurgery, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00102818; 5P50CA190991 (NIH)
Record Dates: First submitted 2022-03-08; First posted 2022-03-16 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Glioma, Malignant
Keywords: ETAPA; Pro00102818; Khasraw; Glioblastoma; Glioma; Duke; Vaccine
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tumor Associated Antigen Peptide Vaccine in Combination with Hiltonol (Experimental): The study vaccine is comprised of three different peptides (small proteins) mixed with Hiltonol®. The three peptides that make up the study vaccine are called pp65, EphA2, and survivin.
  Interventions: Biological: Tumor Associated Antigen Peptide Vaccine P30-EPS Vaccine; Drug: Hiltonol

INTERVENTIONS:
Biological: Tumor Associated Antigen Peptide Vaccine P30-EPS Vaccine — Vaccine that includes 3 peptides (EphA2 linked to P30 peptide, pp65 linked to P30 peptide, and Survivin linked to P30 peptide)
  Other Names: P30-EPS
Drug: Hiltonol — Hiltonol® is made up of synthetic (manmade) RNA (ribonucleic acid) and is used as an adjuvant to the vaccine, meaning it is used with the vaccine to stimulate or enhance the activation of your immune system.
  Other Names: poly-ICLC

SUMMARY:
This is a phase 1b study of P30-linked EphA2, CMV pp65, and survivin vaccination (collectively called the P30-EPS vaccine) in HLA-A*0201 positive patients with a newly diagnosed, unmethylated, and untreated World Health Organization (WHO) grade IV malignant glioma.

DETAILED DESCRIPTION:
This is a phase 1b study of P30-linked EphA2, CMV pp65, and survivin vaccination (collectively called the P30-EPS vaccine) in HLA-A*0201 positive patients with a newly diagnosed, unmethylated, and untreated World Health Organization (WHO) grade IV malignant glioma at the Preston Robert Tisch Brain Tumor Center (PRTBTC) at Duke, is planned to address the following primary objective: Evaluate the safety profile of a cancer vaccine comprised of P30-linked EphA2, CMV pp65, and survivin peptides.

A maximum of 36 patients with a newly diagnosed, previously untreated WHO grade IV malignant glioma that is MGMT promoter unmethylated will be treated in this study after undergoing standard of care surgical resection followed by 6 weeks of radiation therapy (XRT) with concomitant temozolomide (TMZ) and providing informed consent. Patients will receive seven P30 linked-EphA2, -CMV pp65, and -survivin (P30-EPS) peptide vaccines over two phases. The first 5 will be given during the Priming Phase (day 1 through day 22). The final 2 will be given during the Booster Phase (day 84 [± 2 days] and day 140 [± 2 days]). During the Booster Phase on Day 84, patients will also be given 20ug/kg Hiltonol® injections to administer at home every 2 weeks until they return on Day 140. Blood will be drawn throughout the study to investigate the immune response to P30-EPS vaccination. The study will enroll two patient strata: patients who are CMV seronegative and patients who are CMV seropositive. Within each stratum, cohorts of 3 patients will initially be accrued to the study to assess the toxicity associated with the vaccine. The starting dose of P30-EPS is 300 μg/peptide/dose, and the dose will be escalated to 400 μg/peptide/dose. In the event of unacceptable dose-limiting toxicity, the dose will be de-escalated to 200 μg/peptide/dose (dose level minus one). Acute toxicity monitoring will focus on dose-limiting toxicities, as defined in Section 9.1.2 of the protocol, occurring between vaccine 1 and 30 days after vaccine 5. The most common side effects of peptide vaccines are redness or swelling at the injection site, local changes to the texture of your skin (hardening) at the injection site, itching, allergic reactions, and a potentially serious side effect called cytokine release syndrome. The most common side effects of Hiltonol® are reactions at the injection site and flu-like symptoms.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years of age
2. Newly diagnosed Isocitrate dehydrogenase (IDH) wild type (CARIS result), MGMT promoter unmethylated (CARIS result) WHO grade IV glioma (e.g., glioblastoma (GBM) or high grade glioma with molecular features of GBM) with definitive resection prior to enrollment, and residual radiographic contrast enhancement on immediate post-surgical computed tomography (CT), or magnetic resonance imaging (MRI).
3. CMV positive or negative by IgG testing.
4. Karnofsky Performance Status (KPS) of > 70%.
5. Hemoglobin ≥ 9.0 g/dl, absolute neutrophil count (ANC) ≥ 1,000 cells/µl, platelets ≥ 100,000 cells/µl.
6. Serum creatinine ≤ 3 x the upper limit of normal (ULN), serum glutamic oxaloacetic transaminase (SGOT)≤ 3 times ULN
7. Bilirubin ≤ 1.5 times ULN (Exception: Patient has known Gilbert's Syndrome or patient has suspected Gilbert's Syndrome, for which additional lab testing of direct and/or indirect bilirubin supports this diagnosis. In these instances, a total bilirubin of ≤ 3.0 x ULN is acceptable.)
8. Signed informed consent approved by the Institutional Review Board.
9. Female patients must not be pregnant or breast-feeding. Female patients of childbearing potential (defined as < 2 years after last menstruation or not surgically sterile) must use a highly effective contraceptive method (allowed methods of birth control, [i.e. with a failure rate of < 1% per year] are implants, injectables, combined oral contraceptives, intra-uterine device [IUD; only hormonal], sexual abstinence or vasectomized partner) during the trial and for a period of > 6 months following the last administration of trial drug(s). Female patients with an intact uterus (unless amenorrhea for the last 24 months) must have a negative serum pregnancy test within 48 hours prior to first vaccination.
10. Fertile male patients must agree to use a highly effective contraceptive method (allowed methods of birth control [i.e. with a failure rate of < 1% per year] include a female partner using implants, injectables, combined oral contraceptives, IUDs [only hormonal], sexual abstinence or prior vasectomy) during the trial and for a period of > 6 months following the last administration of trial drug(s).

Exclusion Criteria

1. Patients with known potentially anaphylactic allergic reactions to gadolinium-diethylenetriaminepentaacetic acid (DTPA), or any component of the tetanus-diphtheria vaccine.
2. Patients with evidence of tumor in the brainstem, cerebellum, or spinal cord, radiological evidence of multifocal disease, or leptomeningeal disease.
3. Areas of high-grade glioma outside the original radiation field on the post XRT/TMZ MRI.
4. Patients who cannot undergo MRI.
5. Severe, active comorbidity, including any of the following:

   * Unstable angina and/or congestive heart failure requiring hospitalization;
   * Transmural myocardial infarction within the last 6 months;
   * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of first -vaccination;
   * Active infection requiring intravenous treatment or having an unexplained febrile illness (Tmax > 99.5°F/37.5°C)
   * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy;
   * Known hepatic insufficiency resulting in clinical jaundice and/or coagulation defects;
   * Known immunosuppressive disease or Human Immunodeficiency Virus (HIV) and -Hepatitis C positive status;
   * Major medical illnesses or psychiatric impairments that, in the investigator's opinion, will prevent administration or completion of protocol therapy;
   * Active connective tissue disorders, such as lupus or scleroderma that, in the opinion of the treating physician, may put the patient at high risk for radiation toxicity.
6. Co-medication that may interfere with study results (e.g., immuno-suppressive agents other than corticosteroids).
7. Prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin. (Treatment with tamoxifen or aromatase inhibitors or other hormonal therapy that may be indicated in prevention of prior cancer disease recurrence, are not considered current active treatment.)
8. Patients are not permitted to have had any other conventional therapeutic intervention other than surgery, steroids, and standard of care chemoradiation prior to enrollment.
9. Patients who received previous inguinal lymph node dissection or had radiosurgery, brachytherapy, or radiolabeled monoclonal antibodies to treat a CNS tumor will be excluded.
10. Current, recent (within 4 weeks of the administration of this study agent), or planned participation in an experimental drug study.
11. Known history of autoimmune disease (with the exceptions of medically-controlled hypothyroidism and Diabetes Mellitus).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who experience dose-limiting toxicity | 2 months
  Percentage of patients who experience dose-limiting toxicity within each stratum at each dose level

SECONDARY OUTCOMES:
Change in mean fold increase in pp56-specific T cells; Time Frame: Day 1, 22, 84 | 3 months
  Stratified between CMV seropositive and seronegative patients
Change in mean fold increase in EphA2- or survivin- specific T cells; Time Frame: Days 1, 22, 84 | 3 Months
  Amongst all patients
Change in mean fold increase in pp56-specific T cells; Time Frame: Day 1, 22, 84 | 5 months
  Stratified between CMV seropositive and seronegative patients
Change in mean fold increase in EphA2- or survivin- specific T cells; Time Frame: Days 1, 22, 84 | 5 months
  Amongst all patients
Median survival | 36 months
  Amongst all patients
Median progression-free survival | 36 months
  Amongst all patients

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Khasraw, MBChB, MD, FRCP, FRACP, Principal Investigator — Duke University
Locations (1):
- The Preston Robert Tisch Brain Tumor Center at Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Center at Duke University — https://tischbraintumorcenter.duke.edu/
- See also: Duke Health — http://www.dukehealth.org/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2024-12-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT05283109/ICF_000.pdf